CLINICAL TRIAL: NCT03939065
Title: Sensor Augmented Pump (SAP) Therapy for Inpatient Cystic Fibrosis Related Diabetes (CFRD) Management
Brief Title: Sensor Augmented Pump (SAP) Therapy for Inpatient CFRD Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decreased admissions secondary to wider introduction of HEMTs along with pandemic impacted ability to enroll
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-2602
Record Dates: First submitted 2019-04-02; First posted 2019-05-06 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis-related Diabetes; Cystic Fibrosis Pulmonary Exacerbation; Cystic Fibrosis in Children
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Insulin Pump and CGM (Experimental)
  Interventions: Device: Sensor Augmented Pump Therapy
- Standard of Care and CGM (Other)
  Interventions: Device: Standard of Care with CGM

INTERVENTIONS:
Device: Sensor Augmented Pump Therapy — Incorporating both insulin pump and CGM technology together (also known as SAP therapy) has the potential to better optimize glycemic control than each device alone. Participants in this arm will receive their insulin dosing via insulin pump and their blood sugars will be monitored using a Continuous Glucose Monitor.
  Arms: Insulin Pump and CGM
Device: Standard of Care with CGM — Participants assigned to this arm will receive conventional diabetes management with daily insulin injections (or on an insulin pump if already on an insulin pump in the outpatient setting) and capillary blood glucose monitoring. These participants will also wear a blinded Continuous Glucose Monitor (CGM) for outcome assessment.
  Arms: Standard of Care and CGM

SUMMARY:
This research proposes a pilot study using the combination of continuous glucose monitor (CGM) and insulin pump therapy, also known as sensor augmented pump (SAP) therapy, for cystic fibrosis related diabetes (CFRD) management in the inpatient setting, with the aim of improving glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥8 years
2. Confirmed diagnosis of CF by consensus guidelines [50]
3. Diagnosis of CFRD based on American Diabetes Association and CFF criteria [51]
4. Admission for pulmonary exacerbation

Exclusion Criteria:

1. Known type 1 or type 2 diabetes, monogenic diabetes (MODY)
2. Critical illness requiring admission to the intensive care unit
3. Admission for indications other than pulmonary exacerbation (ex. Distal intestinal obstructive syndrome, surgery)
4. Pregnancy

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Differences in CGM percent time over 140 mg/dl | through study completion, up to 3 weeks
  Differences in percent time >140 mg/dl on CGM between groups

SECONDARY OUTCOMES:
Change in Pulmonary Function | baseline and 1 week
  Change in Pulmonary Function, FEV1 (percent and L), from admission to 1 week
Circulatory markers of inflammation | baseline and 1 week
  ∆hsCRP and ∆calprotectin from admission to 1 week
Weight change | baseline and 1 week
  Change in weight from admission to 1 week
Statstrip glucose | through study completion, up to 3 weeks
  glucose obtained from bedside glucometer (mg/dl)

OTHER OUTCOMES:
beta-cell function | within 24 hours of admission
  measures to be derived from oral glucose tolerance testing, including insulin and c-peptide area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chan, MD, Principal Investigator — christinel.chan@childrenscolorado.org
Locations (1):
- Children's Hospital Colorado, University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toner A, McCloy A, Dyce P, Nazareth D, Frost F. Continuous glucose monitoring systems for monitoring cystic fibrosis-related diabetes. Cochrane Database Syst Rev. 2021 Nov 29;11(11):CD013755. doi: 10.1002/14651858.CD013755.pub2. PMID 34844283